CLINICAL TRIAL: NCT01761227
Title: The Safety and Efficacy of Fufangdanshen Tablets in Treatment of Mild to Moderate Vascular Dementia: a 24-week, Double Blind, Randomized, Parallel,Placebo Controlled Trial.
Brief Title: Efficacy and Safety of Fufangdanshen Tablets in Mild to Moderate Vascular Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Hutchison Whampoa Guangzhou Baiyunshan Chinese Medicine Company Limited (Industry)
Responsible Party: Principal Investigator, Jinzhou Tian, Vice precident, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFDA2005L01916; SFDA【2008】I919
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Vascular Dementia
Keywords: Vascular dementia; Fufangdanshen Tablets; Randomized Controlled trial; Chinese Medicine
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fufangdanshen Tablets (Experimental): 1 tablets contains contains tanshinoneⅡA 0.67mg , salvianolic acid B 8.2mg, Panax Notoginsenosides R1 0.53mg, ginsenoside Rb1 3.03mg, ginsenoside Rg1 2.73mg, 3 tablets per time, 3 times per day for 24 weeks
  Interventions: Drug: Fufangdanshen Tablets
- Placebo (Placebo Comparator): 3 tablets per time, 3 times per day for 24 weeks. The placebo has similar smile and appearance as the Fufangdanshen Tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fufangdanshen Tablets — 1 tablets contains contains tanshinoneⅡA 0.67mg , salvianolic acid B 8.2mg, Panax Notoginsenosides R1 0.53mg, ginsenoside Rb1 3.03mg, ginsenoside Rg1 2.73mg, 3 tablets per time, 3 times per day for 24 weeks
  Arms: Fufangdanshen Tablets
Drug: Placebo — Placebo for 3 tablets per time, 3 times per day for 24 weeks
  Arms: Placebo

SUMMARY:
Purpose: The purpose of this study is to examine the efficacy and safety of Fufangdanshen Tablets in patients with mild to moderate vascular dementia (VaD).

DETAILED DESCRIPTION:
This multicenter, double-blind, placebo-controlled study will evaluate the safety and effectiveness of Fufangdanshen Tablets in patients with vascular dementia. All patients will initially receive placebo for a 2 weeks period and then will receive Fufangdanshen Tablets or placebo for 6 months. The primary measures of effectiveness include the change from baseline to the end of treatment in the ADAS-cog/11 score (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and the CIBIC-plus score (Clinician's Interview Based Impression of Change - Plus Caregiver Input). Additional measures of effectiveness include the change from baseline to the end of the treatment in the MMSE score (Mini-mental State Examination), the ADL (Ability of Daily Living) score. Safety evaluations (incidence of adverse events, electrocardiograms (ECGs), physical examinations, laboratory tests) will be performed throughout the study. Patients who complete the double-blind portion of the study will be followed up 12 weeks. Effectiveness will be assessed at 12 weeks, 24weeks and 36 weeks. Safety evaluations (incidence of adverse events, ECGs, physical examinations, laboratory tests) will be performed at 12 weeks, 24weeks and 36 weeks of the study. The study hypothesis is that Fufangdanshen Tablets will be effective in the treatment of patients with vascular dementia and will be well tolerated. Double-blind: Fufangdanshen Tablets: 3 tablets per time, 3 times per day, and placebo : 3 tablets per time, 3 times per day. The placebo has similar smile and appearance as the Fufangdanshen Tablets.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients meeting the diagnostic criteria probable VaD established according to the Diagnostic and Statistical Manual of Mental Disorders (fourth edition) （DSM-Ⅳ） and the National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN)were eligible to participate.
* Weighing between 45 to 90 kg;
* The diagnosis had also to be compatible with the findings from a recent (within last 12 months) magnetic resonance image (MRI) of the brain and
* The Hachinski Ischemia Scale (HIS) score>4.
* six months' mild to moderate VaD duration before inclusion.
* Mild-to-moderate dementia (Score of the Mini-Mental State Examination (MMSE) defined as between 11 to 26)
* The Hamilton Depression Scale (HAMD for 17 items) had a score of ≤ 12
* have a consistent informant to accompany them on scheduled visits
* Ability to read, write, communicate, and understand cognitive testing instructions

Exclusion Criteria:

* Neurodegenerative disorders such as Parkinson's disease, with AD and any other secondary types of dementia;
* cognitive impairment resulting from conditions such as acute cerebral trauma, cerebral damage due to a lack of oxygen, vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor
* having significant psychiatric disease, active peptic ulcer, clinically significant liver, kidney or lung disorders, or heart disease
* history of epilepsy, convulsions, drug abuse or alcohol abuse
* history of hypersensitivity to the treatment drugs;
* concomitant drugs with the potential to interfere with cognition;
* administration of other investigational drugs;
* females of child bearing potential without adequate contraception

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of double-blind treatment Clinician's Interview Based Impression of Change - Plus Caregiver Input; Alzheimer Disease Assessment Scale-cognitive subscale | 24 weeks
  Global cognition was assessed with the CIBIC-plus, at baseline (day 1 clinic visit) and at 12-week intervals thereafter until week 24.
Change in cognitive scores: Alzheimer Disease Assessment Scale-cognitive. subscale (ADAS-cog) | 24 weeks
  Cognition was assessed with the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog), at baseline (day 1 clinic visit) and at 12-week intervals thereafter until week 24.

SECONDARY OUTCOMES:
Change in functional scores: Activities of Daily Living (ADL). | 24 weeks
  Functional ability was evaluated with the ADL was evaluated at baseline (day 1 clinic visit), at the mid-study (week 12), and at the endpoint of treatment (week 24).
Change from baseline to the end of double-blind treatment in Mini-mental state examination (MMSE) scores | 24 weeks
  Change in global cognition:Mini-mental state examination at baseline (day 1 clinic visit) and at 12-week intervals thereafter until week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, Ph.D, M.D, Principal Investigator — Dongzhimen Hospital, Beijing; Jing Shi, M.D, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tian J, Shi J, Wei M, Qin R, Ni J, Zhang X, Li T, Wang Y. The efficacy and safety of Fufangdanshen tablets (Radix Salviae miltiorrhizae formula tablets) for mild to moderate vascular dementia: a study protocol for a randomized controlled trial. Trials. 2016 Jun 8;17(1):281. doi: 10.1186/s13063-016-1410-5. PMID 27266867